CLINICAL TRIAL: NCT01131143
Title: An RCT of Provider-to-Patient IVR Calls to Improve Weight Management in CHCs
Brief Title: Trial of Provider-to-Patient Interactive Voice Response (IVR) Calls to Improve Weight Management in Community Health Centers (CHCs)
Acronym: IVR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Kimberly Hemmerlein, Researcher Coodinator, Indiana University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 0902-70
Record Dates: First submitted 2009-09-14; First posted 2010-05-26 (Estimated); Last update posted 2013-04-02 (Estimated); Status verified 2013-03

CONDITIONS: Obesity
Keywords: Urban community centers; Obesity; Obesity counseling; Low-cost intervention
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Treatment Group 1 (Experimental): Patients will receive a pre-visit, post-referral and post-contact phone call using providers voice
  Interventions: Behavioral: Provider Voice
- Treatment Group 2 (Experimental): Patients will receive a previsit, post-referral and post-contact call using a generic voice
  Interventions: Behavioral: Generic Voice
- Treatment Group 3 (No Intervention): Patients will be provided usual care with no additional phone calls.

INTERVENTIONS:
Behavioral: Provider Voice — A phone call with the pre-recorded doctor's voice will be made to their patients who have been pre-screened for obesity before the patient's appointments prompting the patients to ask about physical activity, nutrition, and weight loss.
  Arms: Treatment Group 1
Behavioral: Generic Voice — A phone call with a pre-recorded neutral voice will be made to the doctor's patients who have been prescreened for obesity before their patient's appointments. The call will prompt them to ask ask their doctor about physical activity, nutrition, and weight loss.
  Arms: Treatment Group 2

SUMMARY:
This study will test the effect of provider to patient interactive voice response (IVR) calls in local Community Health Centers within a weight management program.

DETAILED DESCRIPTION:
We will randomize providers to three groups. Patients whose provider has been randomized to usual care will not receive IVR calls but do have available a guideline-level weight management service in TCL. Groups one and two will receive pre-visit and post-referral calls. The pre-visit call will invite patients who want to discuss weight at their upcoming visit with their provider to remember to do so. The post-referral call will remind patients that they have received a referral and encourage them to schedule a visit with the community based weight intervention program. Patients whose provider has been randomized to group 1 will receive IVR calls using their scheduled and referring provider's voice. Group 2 will receive IVR calls using a standard IVR voice.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients who have screened positive for overweight or obesity

Exclusion Criteria:

* Patients who have not screened positive for overweight or obesity

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1228 (Actual)
Dates: Start 2009-06; Primary Completion 2010-12 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Weight loss refer by provider | 6 months

SECONDARY OUTCOMES:
attendance at program, weight loss | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Daniel O Clark, PhD, Principal Investigator — Indiana School of Medicine
Locations (1):
- Indiana University Center on Aging Research-Regenstrief Institute, Indianapolis, Indiana, United States